CLINICAL TRIAL: NCT01373125
Title: Is the Neosquamous Epithelium "Normal" Following Endoscopic Ablation of Dysplastic Barrett's Esophagus?
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other)
Responsible Party: Principal Investigator, Nicholas Shaheen, MD, Professor of Medicine and Epidemiology Director, Center for Esophageal Diseases and Swallowing, University of North Carolina, Chapel Hill
Other Study IDs: 10-1951
Record Dates: First submitted 2011-06-09; First posted 2011-06-14 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Barrett's Esophagus; Intestinal Metaplasia; Gastroesophageal Reflux Disease (GERD)
Keywords: Barrett's Esophagus; Intestinal metaplasia; Gastroesophageal reflux disease (GERD); Neosquamous epithelium; Radiofrequency ablation (RFA)
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — esophageal biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Radiofrequency Ablation (RFA): Participants in this group are greater than or equal to 12 months status post radiofrequency ablation (RFA).
- Radiofrequency Ablation Longitudinal (RFAL): Participants in this group are part of a longitudinal portion of the study and are enrolled prior to their first radiofrequency ablation procedure and followed at 6 and 12 months after completion of RFA.
- Gastroesophageal Reflux Disease (GERD): Participants in this group have been diagnosed with gastroesophageal reflux disease.
- Asymptomatic Controls (AC): Participants in this group are asymptomatic controls and enrolled as part of the comparison group.

SUMMARY:
The investigators propose a study comparing the morphological and functional aspects of the neosquamous epithelium (NSE) after ablative therapy for dysplastic Barrett's esophagus (BE) to that of native squamous epithelium in normal controls as well as gastroesophageal reflux disease (GERD), non-Barrett's Esophagus (BE) subjects.

DETAILED DESCRIPTION:
Purpose: We propose a study comparing the morphological and functional aspects of the neosquamous epithelium (NSE) after ablative therapy for dysplastic Barrett's esophagus (BE) to that of native squamous epithelium in normal controls as well as gastroesophageal reflux disease (GERD), non-BE subjects.

Participants: Eligible subjects will be women and men between the ages of 18-80, with one of the following:

1. Two or greater cm of dysplastic BE, who will undergo or have undergone radiofrequency ablation for BE at UNC, or
2. Diagnosed with GERD per a gastrointestinal (GI) physician undergoing upper endoscopy for other indications at UNC, or
3. Non-GERD controls per a GI physician with normal esophageal mucosa undergoing upper endoscopy for other indications at UNC.

Procedures (methods): Esophageal biopsies will be obtained specifically for research purposes before ablation therapy or, in subjects not receiving ablative therapy, after completion of the clinically indicated procedure and before withdrawal of the endoscope. Information from the medical record or from patient interview will be obtained regarding diagnosis (Barrett's esophagus, GERD, etc), and a questionnaire administered regarding the duration and frequency of reflux symptoms and complications of reflux disease. Subjects who are enrolled in the pre-ablation group will have additional biopsies and questionnaires administered during scheduled follow-up visits. On the last follow-up visit, this group will also undergo impedance-pH testing using standard methods, to assess for degree of control of esophageal acid exposure, and for number, duration and symptom correlation of non-acid reflux events.

ELIGIBILITY:
Inclusion:

Eligible subjects will be mentally competent women and men between the ages of 18-80, able to speak and read English and who meet one of the following criteria:

* Two or greater cm of dysplastic Barrett's Esophagus (BE), who will undergo or have undergone radiofrequency ablation (RFA) for BE at the University of North Carolina, Chapel Hill (UNC), or
* Diagnosed with gastroesophageal reflux disease (GERD) per a GI physician undergoing upper endoscopy (EGD) for other indications at UNC, or
* Non-GERD controls per a GI physician with normal esophageal mucosa undergoing upper endoscopy for other indications at UNC.

Exclusion:

* Subjects with a bleeding diathesis or other contraindication of endoscopic biopsy.
* Current use of warfarin, heparin, and/or low molecular weight heparin (requires discontinuation of medication 5 days prior to and 7 days after EGD).
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be identified by their gastrointestinal (GI) physician and approached by a study coordinator, nurse, or their GI physician regarding this study on the day of their scheduled procedure at UNC hospitals/GI clinic.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2011-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To characterize reflux symptomatology before and after radiofrequency ablation in subjects with dysplastic Barrett's Esophagus (BE). | Enrollment
  To characterize reflux symptomatology before and after radiofrequency ablation in subjects with dysplastic BE. We will compare before and after gastroesophageal reflux disease (GERD) symptom assessment scale (GSAS) symptom scores using paired Student's t tests. As an exploratory analysis, we will further stratify the data by PPI use (once- vs. twice-daily.

SECONDARY OUTCOMES:
To characterize the physiological and morphological properties of the neosquamous epithelium (NSE) | Enrollment
  To characterize the physiological and morphological properties of the NSE, compared to native esophageal squamous epithelium in healthy controls and subjects with non-Barrett's Esophagus (BE) gastroesophageal reflux disease (GERD). We will compare the physiologic measures of NSE (intercellular space, total electrical resistance (RT), and fluorescein flux) to positive and negative controls using χ2 and Student's t tests.
Correlate the physiologic and morphologic changes in the neosquamous epithelium (NSE) after ablation with the frequency and type of refluxate seen on pH-Impedance. | Enrollment
  We will initially plot esophageal acid exposure (total time with esophageal pH<4) against intercellular space, total electrical resistance (RT), fluorescein flux and gastroesophageal reflux disease (GERD) sysmptom assessment scale (GSAS) scores. R values will be generated. Regression models using each of the 3 physiologic measures (RT, fluorescein, and intercellular space) as the response variable, and acid exposure and number of non-acid reflux events as predictor variables will be generated to define the relationship between reflux type and findings.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Shaheen, MD, MPH, Principal Investigator — UNC-Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States